CLINICAL TRIAL: NCT05697523
Title: Comparison of Respiratory, Physical Activity and Functional Capacities of Patients wıth Mild Relapsing Remitting Multiple Sclerosis and Healthy Controls
Brief Title: Multiple Sclerosis and Respiratory and Functional Capacity
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Principal Investigator, Gürkan Demirtas, Lecturer, Nigde Omer Halisdemir University
Other Study IDs: 60116787-020/92286
Record Dates: First submitted 2023-01-12; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; functional capacity; physical activity; respiratory system; Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: people with mild RRMS
  Interventions: Other: Expanded Disability Status Scale, pulmonary function test, International Physical Activity Questionnaire - Short Form, 6 minute walk test
- Healthy group: healthy people
  Interventions: Other: Expanded Disability Status Scale, pulmonary function test, International Physical Activity Questionnaire - Short Form, 6 minute walk test

INTERVENTIONS:
Other: Expanded Disability Status Scale, pulmonary function test, International Physical Activity Questionnaire - Short Form, 6 minute walk test — Expanded Disability Status Scale, pulmonary function test, International Physical Activity Questionnaire - Short Form, 6 minute walk test

SUMMARY:
It is known that respiratory functions, physical activities and functional capacities of Multiple Sclerosis (MS) patients decrease with the progression of the disease. However, there is not enough information about the severity of the effects of these parameters in mild Relapsing-Remitting Multiple Sclerosis (RRMS) patients. Our aim in this study is to compare the respiratory functions, physical activities and functional capacities of mild RRMS patients with healthy controls and to examine the relationship between them.

DETAILED DESCRIPTION:
It is known that respiratory functions, physical activities and functional capacities of Multiple Sclerosis (MS) patients decrease with the progression of the disease. However, there is not enough information about the severity of the effects of these parameters in mild Relapsing-Remitting Multiple Sclerosis (RRMS) patients. Our aim in this study is to compare the respiratory functions, physical activities and functional capacities of mild RRMS patients with healthy controls and to examine the relationship between them.

Forty individuals diagnosed with RRMS between the ages of 18-60 and 40 healthy individuals with similar demographic characteristics were included in the study.

ELIGIBILITY:
Patient group - Inclusion Criteria:

* Having a definitive diagnosis of RRMS according to the 2017 McDonald criteria
* Being between the ages of 18-60.
* To be willing to participate in the study.
* EDSS score between 0-3.

Healthy group - Inclusion Criteria:

* Being between the ages of 18-60.
* To be willing to participate in the study.

Patient group - Exclusion Criteria:

* Have other neurological, orthopedic and systemic problems
* Having a relapse 30 days before or during the study
* Changes in medication use in the past 30 days

Healthy group - Exclusion Criteria:

* Have neurological, orthopedic and systemic problems

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Multiple Sclerosis patients who applied to Pamukkale University Hospital Neurology Clinic were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function Tests- FEV1/FVC | Baseline
  Evaluation of FEV1/FVC ratio MicroQuark® computer-based USB spirometer will be used to assess the respiratory function of the participants. The person will be asked to take a few normal breaths followed by as deep a breath as possible and instructed to exhale forcefully and quickly without waiting. The test will be terminated by instructing the participant to take a deep breath after exhaling for at least six seconds.
Pulmonary Function Tests- FVC | Baseline
  Evaluation of Forced Vital Capacity (FVC) MicroQuark® computer-based USB spirometer will be used for FVC evaluation. The person will be asked to take a few normal breaths, then take as deep a breath as possible, and then exhale forcefully and quickly without waiting. The test will be terminated by instructing the participant to take a deep breath after exhaling for at least six seconds.
Pulmonary Function Tests- FEV1 | Baseline
  Evaluation of Forced Expiratory Volume in 1 second (FEV1) MicroQuark® computer-based USB spirometer will be used for FEV1 evaluation. The person will be asked to take a few normal breaths, then take as deep a breath as possible, and then exhale forcefully and quickly without waiting. The test will be terminated by instructing the participant to take a deep breath after exhaling for at least six seconds.
Pulmonary Function Tests- PEF | Baseline
  Evaluation of Peak Expiratory Flow (PEF) MicroQuark® computer-based USB spirometer will be used for PEF evaluation. The person will be asked to take a few normal breaths, then take as deep a breath as possible, and then exhale forcefully and quickly without waiting. The test will be terminated by instructing the participant to take a deep breath after exhaling for at least six seconds.
Pulmonary Function Tests- MVV | Baseline
  Maximum voluntary ventilation (MVV) MicroQuark® computer-based USB spirometer will be used for MVV evaluation. Then the participant will take the disposable bacteria filter mouthpiece between his lips and holds it tightly. The person will be asked to deeply and rapidly breaths for 10 to 15 seconds.
Functional Capacity | Baseline
  The 6-minute walk test (6MWT) was used to measure functional capacity. In the test, the participant was asked to walk for 6 minutes as fast as possible in a 30-meter corridor, and the total distance in meters was recorded. Standard encouragement was given to the participant every 60 seconds during the test. Estimated values of participants For men; (7.57 x height(cm)) - (5.02 x age) - (1.76 x kg) - 309, for women; Calculated with the formula (2.11 x height(cm)) - (2.29 x kg) - (5.78 x age) + 667.
International Physical Activity Questionnaire - Short Form | Baseline
  The International Physical Activity Questionnaire-Short Form (IPAQ-SF) was used to evaluate physical activity. It was developed to evaluate the physical activities of people between the ages of 15-60 in their daily lives. It consists of seven questions in total and questions the time spent in vigorous, moderate-to-severe and walking activities. In addition, the sitting time is considered as a separate question. The Metabolic Equivalent (MET-minute) score is determined at the end of the calculation made by multiplying the MET value of the activities performed by the minute. Classification is based on the numerical data obtained. Accordingly, there are 3 activity levels: Inactive, minimal active and very active. The lowest level of physical activity is inactive and the highest level of physical activity is very active. The IPAQ is a valid and reliable test in MS patients.

SECONDARY OUTCOMES:
Expanded Disability Status Scale | Baseline
  The Expanded Disability Status Scale is a method of quantifying disability in multiple sclerosis. The scale is based on a neurological examination by a clinician. It has steps from 0 to 10. The higher scores indicate higher neurological disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No